CLINICAL TRIAL: NCT06519968
Title: A Single-blind, Randomised, Placebo-controlled Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Inhaled AZD4604 Following Single Ascending and Multiple Doses in Healthy Japanese and Chinese Participants
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Inhaled AZD4604 in Healthy Japanese and Chinese Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D8210C00002
Record Dates: First submitted 2024-07-05; First posted 2024-07-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: Ascending doses; Multiple doses; JAK1 inhibitor; Chinese; Japanese

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part 1a: AZD4604 (Dose 1) SAD (Experimental): Japanese participants will receive single dose of AZD4604 (Dose 1) via inhalation on Day 1.
  Interventions: Drug: AZD4604
- Part 1a: AZD4604 (Dose 2) SAD (Experimental): Japanese participants will receive single dose of AZD4604 (Dose 2) via inhalation on Day 1.
  Interventions: Drug: AZD4604
- Part 1a: AZD4604 (Dose 3) SAD (Experimental): Japanese participants will receive single dose of AZD4604 (Dose 3) via inhalation on Day 1.
  Interventions: Drug: AZD4604
- Part 1a: Placebo (Placebo Comparator): Japanese participants will receive single dose of matching placebo to AZD4604 on Day 1.
  Interventions: Drug: Placebo
- Part 1b: AZD4604 (Dose 4) Multiple dose cohort (Experimental): Japanese participants will receive AZD4604 (Dose 4) via inhalation twice daily (BID) from Day 1 to Day 6 and a single dose on Day 7.
  Interventions: Drug: AZD4604
- Part 1b: Placebo (Placebo Comparator): Japanese participants will receive matching placebo to AZD4604 BID from day 1 to day 6 and a single dose of placebo on Day 7.
  Interventions: Drug: Placebo
- Part 2a: AZD4604 (Dose 1) SAD (Experimental): Chinese participants will receive single dose of AZD4604 (Dose 1) via inhalation on Day 1.
  Interventions: Drug: AZD4604
- Part 2a: AZD4604 (Dose 3) SAD (Experimental): Chinese participants will receive single dose of AZD4604 (Dose 3) via inhalation on Day 1.
  Interventions: Drug: AZD4604
- Part 2a: Placebo (Placebo Comparator): Chinese participants will receive single dose of matching placebo to AZD4604 on Day 1.
  Interventions: Drug: Placebo
- Part 2 b: AZD4604 (Dose 4) Multiple dose cohort (Experimental): Chinese participants will receive AZD4604 (Dose 4) via inhalation BID from Day 1 to Day 6 and a single dose on Day 7.
  Interventions: Drug: AZD4604
- Part 2b: Placebo (Placebo Comparator): Chinese participants will receive placebo via inhalation BID from Day 1 to Day 6 and a single dose on Day 7.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4604 — AZD4604 will be administered as Dry Powder Inhalation (DPI).
  Arms: Part 1a: AZD4604 (Dose 1) SAD; Part 1a: AZD4604 (Dose 2) SAD; Part 1a: AZD4604 (Dose 3) SAD; Part 1b: AZD4604 (Dose 4) Multiple dose cohort; Part 2 b: AZD4604 (Dose 4) Multiple dose cohort; Part 2a: AZD4604 (Dose 1) SAD; Part 2a: AZD4604 (Dose 3) SAD
Drug: Placebo — Placebo will be administered as DPI.
  Arms: Part 1a: Placebo; Part 1b: Placebo; Part 2a: Placebo; Part 2b: Placebo

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, and pharmacokinetics (PK) of AZD4604 when administered as single or multiple inhaled doses to healthy Japanese and Chinese participants.

DETAILED DESCRIPTION:
This study will comprise of two parts: Part 1 and Part 2

Part 1 will investigate the safety, tolerability, and PK of inhaled AZD4604 following single ascending and multiple doses in healthy Japanese participants.

Part 1a will include three single ascending dose (SAD) cohorts and Part 1b will include one multiple dose cohort.

Part 2 will investigate the safety, tolerability, and PK of inhaled AZD4604 following single ascending and multiple doses in healthy Chinese participants.

Part 2a will include two SAD cohort and Part 2b will include one multiple dose cohort.

Part 1a and Part 2a will comprise of:

1. A Screening Visit within 28 days before dosing.
2. A treatment period (Day 1 to Day 7)
3. A final assessment on Day 7

Part 1b and Part 2b will comprise of:

1. A Screening Visit within 28 days before dosing.
2. A treatment period (Day 1 to Day 13)
3. A final assessment on Day 13

ELIGIBILITY:
Inclusion Criteria:

* Japanese participants who are born in Japan, has 2 Japanese biological parents, 4 Japanese grandparents as confirmed by the interview and has lived outside Japan for less than 10 years at the time of screening.
* Chinese participants who are born in China, has 2 Chinese biological parents, 4 Chinese grandparents as confirmed by the interview and has lived outside China for less than 10 years at the time of screening.
* Have body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 45 kg.
* Healthy participants must have a Forced Expiratory Volume at first breath (FEV1) ≥ 80% of the predicted value in accordance with American Thoracic Society (ATS)/European Respiratory Society (ERS) criteria at the Screening and admission visits.
* Female participants must have a negative pregnancy test.

Exclusion Criteria:

* History or presence of clinically important disease which may put participant at risk because of participation in study.
* Participant has an increased risk of infection.
* History of malignancy other than superficial basal cell carcinoma, having a first degree relative with lung cancer or disease history suggesting abnormal immune function.
* Has received any vaccine 30 days prior to first dose.
* Has a body temperature of > 37.7°C on Day -1.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Known or suspected history of drug abuse, alcohol abuse or excessive intake of alcohol.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes, vaping, and nicotine replacement therapy) within the previous 6 months or has a smoking history of > 5 pack-years.
* History of a serious or severe adverse reaction to AZD4604 or any of its additive constituents.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4604.
* Plasma donation within 1 month of the Screening Visit or any blood donation/blood loss> 500 mL during the 3 months prior to the Screening Visit.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12-lead safety ECG.
* Female participants who are planning a pregnancy during the study period or within 1 month after the last dose of study intervention.
* Abnormal vital signs at the Screening Visit, after 5 minutes supine rest.
* History of any significant respiratory disorders such as asthma (a history of childhood asthma without symptoms or treatment after the age of 10 years is allowable), chronic obstructive pulmonary disease, or idiopathic pulmonary fibrosis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse event (AEs) | From Day -28 to 5 weeks (Parts 1a and 2a); Day -28 to 6 weeks (Parts 1b and 2b)
  To assess the safety and tolerability of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).

SECONDARY OUTCOMES:
Maximum observed plasma (peak) drug concentration (Cmax) | From Day 1 to Day 7 (Parts 1a and 2a); From Day 1 to Day 13 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).
Time to reach peak or maximum observed concentration following drug administration (tmax) | From Day 1 to Day 7 (Parts 1a and 2a); From Day 1 to Day 13 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).
Terminal elimination rate constant (λz) | From Day 1 to Day 7 (Parts 1a and 2a); From Day 1 to Day 13 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).
Half-life associated with terminal slope of a semi-logarithmic concentration time curve (t½λz) | From Day 1 to Day 7 (Parts 1a and 2a); From Day 1 to Day 13 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).
Partial area under concentration-time curve from time 0 to 12 hours (AUC [0-12]) | From Day 1 to Day 7 (Parts 1a and 2a); On Day 1 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).
Partial area under concentration-time curve from time 0 to 24 hours (AUC [0-24]) | From Day 1 to Day 7 (Parts 1a and 2a); From Day 1 to Day 13 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).
Area under the plasma concentration curve from zero to last quantifiable concentration (AUClast) | From Day 1 to Day 7 (Parts 1a and 2a); From Day 1 to Day 13 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).
Area under the plasma concentration curve from zero to infinity (AUCinf) | From Day 1 to Day 7 (Parts 1a and 2a)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a).
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | From Day 1 to Day 7 (Parts 1a and 2a); From Day 1 to Day 13 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).
Volume of distribution (apparent) at steady state following extravascular administration based on terminal phase (Vz/F) | From Day 1 to Day 7 (Parts 1a and 2a); From Day 1 to Day 13 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).
Area under the plasma concentration time curve from zero to the last quantifiable concentration, divided by dose (AUClast/D) | From Day 1 to Day 7 (Parts 1a and 2a); From Day 1 to Day 13 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).
Area under the plasma concentration curve from zero to infinity, divided by dose (AUCinf/D) | From Day 1 to Day 7 (Parts 1a and 2a)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a).
Maximum observed plasma (peak) drug concentration, by dose (Cmax/D) | From Day 1 to Day 7 (Parts 1a and 2a); From Day 1 to Day 13 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).
The last time point at which the concentration is measured (tlast) | From Day 1 to Day 7 (Parts 1a and 2a); From Day 1 to Day 13 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as single ascending doses (Parts 1a and 2a), and multiple doses (Parts 1b and 2b).
Area under plasma concentration time curve from zero to end of dosing interval (AUCτ) | From Day 1 to Day 13 (Parts 1b and 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as multiple doses (Parts 1b and 2b).
Area under plasma concentration time curve from zero to end of dosing interval, by dose (AUCτ/D) | From Day 1 to Day 13 (Parts 1b to 2b)
  To characterise the plasma PK of AZD4604 following inhaled administration of AZD4604 as multiple doses (Parts 1b and 2b).
Cough Severity self-assessment as measured by Visual Analogue Scale (VAS) | From Day 1 to Day 8 (Parts 1b and 2b)
  The cough VAS is a brief and simple measure of cough severity. It consists of a 100 mm vertical scale on which the participant is asked to place a cross at the point that indicates the severity of his/her cough in the last 24 hours between "No cough" and "Worst cough ever". The position of the cross is measured from the "No cough" reference point. A minimal clinically important difference is considered to be a 17 mm change from previous.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: D8210C00002_CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8210C00002&attachmentIdentifier=6a80ec34-ffbf-4328-9e7c-0ab2e2790948&fileName=D8210C00002_CSR_Synopsis+CSR_Errata_Redacted.pdf&versionIdentifier=
- See also: Astrazenecaclinicaltrials.com-study results — https://www.astrazenecaclinicaltrials.com/study/D8210C00002/